CLINICAL TRIAL: NCT05794568
Title: Multicenter, Open, Controlled, Randomized Study to Evaluate the Efficacy of the OITcontrol Application in Monitoring Patients in OIT With Food.
Brief Title: Evaluate the Efficacy of the OITcontrol Application.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OITcontrol_QL
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2022-11

CONDITIONS: Food Allergy in Children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OITcontrol group (Active Comparator)
  Interventions: Device: OITcontrol app monitoring
- paperPRO group (No Intervention)

INTERVENTIONS:
Device: OITcontrol app monitoring — App to monitor OIT patients
  Arms: OITcontrol group

SUMMARY:
The main aim of this study is to evaluate the clinical efficacy of the OITcontrol application in patients undergoing OIT of eggs or milk used during the follow-up of this treatment.

DETAILED DESCRIPTION:
1. Evaluate the quality of life of patients with respect to their food allergy by analyzing the data from the FAQLQ-CF and/or SFAQoL-PF questionnaires.
2. Evaluate the perception of patients on the quality and safety of hospital care through the analysis of the adapted SERVQHOS questionnaire and the "Evolution of the perception of patients on the safety of health services".
3. Evaluate patient safety with OITcontrol based on:

   1. Number of reactions in the hospital,
   2. Number of reactions outside the hospital,
   3. Compliance with the information and recommendations by the patient:

   i. recording shots, ii. reaction log, iii. discordances between the medication used and prescribed after a reaction, iv. avoidance of cofactors.
4. Evaluate the consumption of health resources regarding the use, derived from the OIT of the following resources:

   1. Number of extraordinary visits to the allergy department,
   2. Number of phone calls for questions,
   3. Number of visits to the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be between 4 and 12 years old at the time of informed consent.
* Patients diagnosed with food allergy to eggs and/or milk (clinical history compatible with IgE-mediated reaction with egg or milk together with positive specific IgE against egg white or milk (>0.35kU/L) and/or skin test by intraepidermal puncture equal to or similar to 3mm for egg white or milk); in case of egg allergy, patients may be allergic to raw or undercooked egg despite their tolerance to well-cooked egg.
* The patient, or their legally authorized representative, has given their consent to participate in the study.
* The patient, or his legally authorized representative, has accepted the OIT treatment after the explanation of its risks and benefits and the requirements for the maintenance phase.
* The patient must, in the opinion of the investigator, be able to meet all the requirements of the study.
* The patient, or their legally authorized representative, who assumes the OIT treatment at home, has a Smartphone with internet access via mobile data and/or Wi-Fi available at home.
* Reaction with the OIT allergen in the controlled oral provocation test (POC) included in the initial phase of treatment.

Exclusion Criteria:

* Present any of the OIT exclusion criteria:

  1. Allergy to cow's milk and/or eggs not mediated by IgE.
  2. Uncontrolled asthma. In the case of a patient with asthma, this must be controlled before the start of OIT.
  3. Severe atopic dermatitis.
  4. Previous diagnosis of eosinophilic esogaphitis.
  5. Inflammatory bowel disease.
  6. Mastocytosis.
  7. Immunocompromised patients.
  8. Disorders and/or treatments in which the use of adrenaline is contraindicated.
  9. Difficulty understanding the risks and benefits of the procedure, and social and family factors that may compromise long-term maintenance therapy. This includes conflicts between parents or legal representatives that may adversely affect treatment.
  10. Inability of parents or legal representative to follow instructions, identify reactions, or administer medication (especially auto-injectable adrenaline).
* Previous allergic reaction with the corresponding OIT food within the month prior to the initial visit.
* Treatment with omalizumab or any other immunomodulatory biologic drug within the three months prior to the initial visit.
* Pregnant women, or women of childbearing potential not using a safe means of contraception (abstinence is considered an acceptable method) during the entire study period.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The effectiveness of OITcontrol as an application to improve the quality of life. | 12 weeks
  Improve the quality of life of patients, as well as their perception of the quality and safety of hospital care, safety and the reduction of the consumption of health resources in patients under OITcontrol.
  * Baseline variables of the patient's clinical history in relation to their allergy to the allergen in the OIT, their base treatment and/or premedication, and the baseline sensitization parameters (skin test, total and specific IgE to the allergen of the OIT) obtained in the V0. The variables of the first day of treatment will be collected: threshold dose, last tolerated dose, and type of reaction presented.
  * The variables in the escalation visits will be taken in the space of time between two hospital visits. The data to be collected in a hospital visit correspond to the events that occurred during that hospital visit and in the home doses or extraordinary hospital visits of the previous week from the last ordinary hospi

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Hospital Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Severo Ochoa, Leganés, Madrid
  - Universidad de Navarra, Pamplona, Navarre
  - Hospital Gregorio Marañón, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid